CLINICAL TRIAL: NCT01540409
Title: Open-Label, Multiple-Dose, Efficacy, Safety, and Tolerability Study of Eteplirsen in Subjects With Duchenne Muscular Dystrophy Who Participated in Study 4658-US-201
Brief Title: Efficacy, Safety, and Tolerability Rollover Study of Eteplirsen in Subjects With Duchenne Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4658-us-202
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: DMD, Duchenne, Eteplirsen, dystrophy, dystrophin, exon 51
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVI-4658 (Eteplirsen) (Experimental): Multiple-Dose Extension Study
  Interventions: Drug: AVI-4658 (Eteplirsen)

INTERVENTIONS:
Drug: AVI-4658 (Eteplirsen) — Eteplirsen will be administered once weekly via an IV infusion. There are two treatment groups, 30 mg/kg and 50 mg/kg.
  Other Names: EXONDYS 51

SUMMARY:
The primary objective of this study is to assess the ongoing efficacy, safety, and tolerability of an additional 212 weeks of treatment with eteplirsen injection in Duchenne muscular dystrophy (DMD) subjects who have successfully completed the 28 week eteplirsen study: Study 4658-us-201. This study will also evaluate the correlation between biomarkers for DMD and the clinical status of participating DMD subjects.

DETAILED DESCRIPTION:
This is an open label, multiple dose extension study to assess the ongoing efficacy, safety, and tolerability of weekly intravenous (IV) infusions of eteplirsen in DMD subjects who have successfully completed Study 4658-us 201.

Subjects will have the opportunity to enroll in this study during the last visit of Study 4658-us-201 (Week 28). Eligible subjects will receive once weekly IV infusions of eteplirsen (50 or 30 mg/kg) for an additional 212 weeks. Subjects will receive the same dose of eteplirsen they received in Study 4658-us-201. Subjects will thereafter continue to receive once weekly IV infusions of eteplirsen for up to an additional 72 week period (through week 284). If commercial eteplirsen becomes available during this additional 72 week period, participation in the study will be discontinued as subjects transition to commercial eteplirsen.

Safety, efficacy, pharmacokinetic (PK), and biomarker assessments will be performed at scheduled visits; adverse events (AEs) and concomitant medications and therapies will be continuously monitored.

If review of data from this open label study suggests that continued treatment with eteplirsen is warranted, this study may be extended by protocol amendment or subjects who successfully complete this study may have the opportunity to participate in a separate follow on, open label eteplirsen study.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for this study.

1. The subject and/or their parent/legal guardian are willing and able to provide signed informed consent.
2. The subject has successfully completed 28 weeks of treatment in Study 4658-US-201.
3. The subject has a parent(s) or legal guardian(s) who is able to understand and comply with all of the study procedure requirements.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from this study.

1. The subject has a prior or ongoing medical condition that, in the Investigator's opinion, could adversely affect the safety of the subject or make it unlikely that the course of treatment or follow-up would be completed or impair the assessment of study results.

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (11):
- United States (11):
  - Miller Children's Hospital, Long Beach, California
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University Medical School, St Louis, Missouri
  - Summerwood Pediatrics/Infusacare Medical Services, Liverpool, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Specialty Group, Pediatric Neurology, Norfolk, Virginia
  - Osceola Medical Center, Osceola, Wisconsin

REFERENCES:
- [Derived] Mendell JR, Goemans N, Lowes LP, Alfano LN, Berry K, Shao J, Kaye EM, Mercuri E; Eteplirsen Study Group and Telethon Foundation DMD Italian Network. Longitudinal effect of eteplirsen versus historical control on ambulation in Duchenne muscular dystrophy. Ann Neurol. 2016 Feb;79(2):257-71. doi: 10.1002/ana.24555. Epub 2016 Jan 8. PMID 26573217
- See also: Mendell, 2013, Annals of Neurology — https://www.ncbi.nlm.nih.gov/pubmed/?term=23907995
- See also: Mendell, 2016, Annals of Neurology — https://www.ncbi.nlm.nih.gov/pubmed/?term=26573217
- See also: Kinane, 2018, Journal of Neuromuscular Diseases — https://www.ncbi.nlm.nih.gov/pubmed/?term=Kinane+eteplirsen
- See also: Charleston, 2018, Neurology — https://www.ncbi.nlm.nih.gov/pubmed/29752304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 centers in the United States. Overall, 12 participants who completed parent study 4658-us-201 (NCT01396239) were enrolled between July 2011 and February 2012 in this extension study (4658-us-202; NCT01540409). A 4-week open label period (Week 24-28) was observed between the parent and extension study.
Pre-assignment Details: Participants who received placebo in 4658-us-201 study were randomized in 1:1 ratio in this extension study to receive either eteplirsen 30 or 50 milligram per kilogram (mg/kg) and, those who received eteplirsen 30 or 50 mg/kg in 4658-us-201 received same treatment in this extension study.
Groups:
- Eteplirsen 30 mg/kg: Participants who received 30 milligram per kilogram (mg/kg) eteplirsen or placebo once weekly, intravenous (IV) infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), continued the same treatment with 30 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
- Eteplirsen 50 mg/kg: Participants who received 50 mg/kg eteplirsen or placebo once weekly, IV infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), continued the same treatment with 50 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
Period: Overall Study
Arm/Group | Eteplirsen 30 mg/kg | Eteplirsen 50 mg/kg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized participants who received any amount of study drug.
Groups:
- Eteplirsen 30 mg/kg: Participants who received 30 mg/kg eteplirsen or placebo once weekly, IV infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), continued the same treatment with 30 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
- Total: Total of all reporting groups
Arm/Group | Eteplirsen 30 mg/kg | Eteplirsen 50 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (0.75) | 8.8 (1.47) | 9.0 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 6 Minute Walk Test (6MWT) at Week 240
Description: This study used a modified version of the 6MWT test procedure described in American Thoracic Society (ATS) 2002 guidelines, specifically adapted for patients with Duchenne muscular dystrophy. The participant was asked to walk a set course of 25 meters for 6 minutes (timed) and the distance walked in meters was recorded. Increases from baseline in 6MWT distance are indicative of improvement and decreases from baseline indicate worsening. Baseline here corresponds to the baseline in the parent study (4658-us-201, NCT01396239).
Time Frame: Parent Baseline and Week 240
Population: The Intent-to-Treat Population (ITT) population included all participants randomized into parent study 4658-us-201. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Results are reported below in 2 reporting groups based on evaluation period (Week 240) as applicable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Eteplirsen 30 mg/kg | Eteplirsen 50 mg/kg
Number analyzed (Participants) | 4 | 3
Meters | -199.0 (113.25) | -258.0 (175.65)

2. Primary Outcome: Change From Baseline in the Percentage of Dystrophin Positive Fibers (PDPF) at Week 48
Description: Dystrophin expression as assessed by percent dystrophin positive fibers was measured by immunohistochemistry (IHC) technique using primary anti-dystrophin antibody. Percent change from baseline is the arithmetic difference of the treatment time point minus baseline divided by baseline calculated for individual subjects. Baseline here corresponds to the baseline in the parent study (4658-us-201, NCT01396239).
Time Frame: Parent Baseline and Week 48
Population: The ITT population included all participants randomized into parent study 4658-us-201. Results are reported below in 3 reporting groups of placebo to eteplirsen, eteplirsen 30 mg/kg, and eteplirsen 50 mg/kg, respectively, based on evaluation period (Week 48) as applicable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of Dystrophin Positive Fibers
Groups:
- Placebo to Eteplirsen: Participants who received eteplirsen matched placebo once weekly, IV infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), followed by 30 or 50 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
- Eteplirsen 30 mg/kg: Participants who received 30 mg/kg eteplirsen once weekly, IV infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), continued the same treatment with 30 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
- Eteplirsen 50 mg/kg: Participants who received 50 mg/kg eteplirsen once weekly, IV infusion for 24 weeks in the parent study 4658-us-201 (NCT01396239), continued the same treatment with 50 mg/kg eteplirsen once weekly for 212 weeks (up to Week 240) in this extension study.
Arm/Group | Placebo to Eteplirsen | Eteplirsen 30 mg/kg | Eteplirsen 50 mg/kg
Number analyzed (Participants) | 4 | 4 | 4
Percentage of Dystrophin Positive Fibers | 37.70 (12.602) | 51.69 (7.089) | 42.93 (13.433)

ADVERSE EVENTS:
Time Frame: Parent Baseline up to 240 weeks (cumulative Study 4658-us-201 + 4658-us-202)
Description: Only treatment-emergent adverse events with an onset date on or after the date of first dose of study drug were reported. Relatedness of Serious Adverse Events (SAEs) to study medication was determined by the Investigator.
Arm/Group | Eteplirsen 30 mg/kg | Eteplirsen 50 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=6) | Eteplirsen 50 mg/kg (N=6)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 — Not related to study medication. All events are related to patients falling.
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 1 — Not related to study medication. All events are related to patients falling.
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 0 — Not related to study medication.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Not related to study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eteplirsen 30 mg/kg (N=6) | Eteplirsen 50 mg/kg (N=6)
Procedural pain (Injury, poisoning and procedural complications) | 5 | 6
Contusion (Injury, poisoning and procedural complications) | 4 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 2
Excoriation (Injury, poisoning and procedural complications) | 2 | 3
Joint injury (Injury, poisoning and procedural complications) | 2 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 3
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 4
C-reactive protein increased (Investigations) | 2 | 2
Blood glucose increased (Investigations) | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Body height below normal (Investigations) | 1 | 1
Activated partial thromboplastin time abnormal (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Red blood cells urine positive (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Wound healing normal (Investigations) | 0 | 1
Headache (Nervous system disorders) | 4 | 5
Balance disorder (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 3
Oral pain (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Retained deciduous tooth (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Catheter site pain (General disorders) | 2 | 2
Infusion site extravasation (General disorders) | 2 | 2
Device occlusion (General disorders) | 1 | 1
Infusion site haematoma (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 2 | 0
Thrombosis in device (General disorders) | 2 | 1
Application site erythema (General disorders) | 0 | 1
Application site pruritus (General disorders) | 0 | 1
Catheter site haematoma (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Infusion site pain (General disorders) | 0 | 1
Infusion site rash (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Swelling (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Papule (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria thermal (Skin and subcutaneous tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 2
Hordeolum (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 0 | 3
Post procedural cellulitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 2
Candidiasis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tinea capitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Obesity (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 4
Glycosuria (Renal and urinary disorders) | 0 | 1
Hypercalciuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Cataract subcapsular (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 1
Hypermetropia (Eye disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Goitre (Endocrine disorders) | 0 | 1
Growth hormone deficiency (Endocrine disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Infusion site urticaria (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Paraspinal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Torus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigators and the Sponsor (or its agents) that restricts the PIs' rights to discuss or publish trial results after the trial is completed.